CLINICAL TRIAL: NCT03240653
Title: Predictive Measures to Stratify Clinical Outcomes in Children and Adults With Gaucher Disease and Responses to Specific Therapies
Brief Title: Gaucherite - A Study to Stratify Gaucher Disease
Acronym: Gaucherite
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Timothy Cox MD, Professor of Medicine Emeritus, Director of Research, Honorary Consultant, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: MR/K015338/1
Record Dates: First submitted 2017-07-12; First posted 2017-08-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Gaucher Disease, Type I; Gaucher Disease, Type III
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine, Blood (Plasma, Serum, EDTA) Fresh Tissue, Biopsy, Bone Marrow Aspiration & Cerebro-spinal fluid (rarely).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Type III: Stratified response to EnzymeTherapy Substrate Reduction Therapy (expected) Splenectomy (and interactions)
  Interventions: Other: Stratified response to Enzyme Therapy
- Patients Type I: Stratified response to Enzyme Therapy and Substrate Reduction Therapy- Splenectomy (and interactions)
  Interventions: Other: Stratified response to Enzyme Therapy

INTERVENTIONS:
Other: Stratified response to Enzyme Therapy — Observational study involves review of retrospective and prospective data of participants' medical history, pathology, imaging and health questionnaires.
  Other Names: Stratified response to Substrate Reduction Therapy; Splenectormy

SUMMARY:
The purpose of this research is to review data already collected and to collect new data from adults and children in England with Gaucher Disease to determine clinical factors which predict severity and response to therapy of Gaucher disease especially in the areas of bone, cancer and brain conditions.

DETAILED DESCRIPTION:
Gaucher disease is part of a rare group of genetic metabolic diseases which are caused by an inherited deficiency of the enzyme glucocerebrosidase. The most common form, Type 1 affects 1 in 40,000 to 60,000 individuals in the general population. In Type 1 symptoms may appear at any time from infancy to old age. The disease is associated with anaemia (a decrease in the amount of red blood cells), fatigue (tiredness), bruising and an increased tendency to bleed. An enlarged spleen and liver with stomach swelling may also occur as well as bone pain, fractures and bone deterioration. Type 1 was formerly considered not to affect the brain or nervous system. Some patients with Type 1 Gaucher disease have no symptoms, while others develop serious symptoms that can be life threatening; latterly Parkinsonism and Dementia with Lewy bodies has been noted to occur with increased frequency in patients with this variant of Gaucher disease compared with healthy control subjects in an age-matched population.

In Gaucher Disease Type 3 the brain and spinal cord are affected. Type 3 is rare and affects fewer than 1 in 100,000 people. The brain and spinal cord symptoms in Type 3 are less severe than in those who have evidence of florid neurologocal disease in infancy years of age. The symptoms of the brain and spinal cord appear in early to late childhood, and patients with Type 3 Gaucher disease live often, but not always, well into adulthood.

Gaucher disease is not gender-specific and its signs and symptoms may appear in affected individuals at any age, with Type 3 being commonly diagnosed in childhood. Although individuals from any ethnic background may develop Gaucher disease, Type 1 Gaucher disease is most common among Jews of Ashkenazi (Eastern European) descent. Among this group, about 1 in 900 people are at risk of Gaucher disease.

There are approximately 280 people in England diagnosed with Gaucher Disease, who receive treatment or management at one of the treating hospitals.

Patients with Gaucher disease have an increased risk of developing myeloma and Parkinson's disease. Myeloma, also known as multiple myeloma, is a type of bone marrow cancer affecting the white blood cells of the immune system which generate antibodies. Approximately 1 in 10 Gaucher patients have a specific blood protein - a monoclonal antibody called a paraprotein, which is found in both malignant and non-malignant conditions, including myeloma.

Parkinson disease is a neurological condition which develops over time as specific brain cells that control movement, die. The failure to produce less of a chemical called dopamine, reduces communication between brain cells involved in the coordination of movement, behaviour, learning and memory.

The investigators will collect information from patients diagnosed with Gaucher disease and any of the conditions mentioned above (for which the patient is already being monitored). Further information required about their clinical status will be obtained from their past and on-going medical records; this will be done as the participants attend hospital as part of their routine care for Gaucher disease. The information we need for the research is no different from the information which is already recorded and will be recorded in their medical notes when they come to the hospital for their routine care, every 6 months.

For the purpose of this study, the investigators will take a few extra blood samples from the participant. These samples will be used to conduct biochemical and cellular analysis solely for the purpose of this research.

The Investigators also request permission from participants to allow access and use for the purpose of the research any archived biological material (blood serum and/or tissue) which may be available from the medical procedures that has been received in the past.

In addition, for the purpose of this research, at each visit, investigators request that the participant also completes questionnaires about physical and social abilities, mental health and quality of life.

All the research-specific procedures (i.e. procedures that the participant would not normally receive during their standard of care hospital visits) can be carried out at either their routine clinic appointments or at another time that the participant would find convenient.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this study:

1. Confirmed biochemical diagnosis of Type I, Type II or Type III Gaucher disease
2. Written Ethics Committee (EC) approved informed consent obtained from the patient, or patient's parent or legal guardian and patient assent if appropriate
3. Male or Female patients, no age limitation
4. Willing and able to comply with study schedule and procedures
5. Deceased patients for whom the EC determines that patient data can be collected without a new consent from the patient

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the study:

1. Unrelated co-morbid condition limiting life expectancy to less than 6 months
2. Patient or if applicable, parent or legal guardian is unable to comprehend, sign and date the EC approved informed consent form and patient assent as appropriate
3. If determined unsuitable for the study by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Seven (previously eight) specialized centres for Gaucher disease in England will recruit approximately 280 patients.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome | 2029
  Presence of saccadic ocular deficits
Fragility Fracture | 2029
  Dual energy absorptive photiometry (DEXA) will allow us to measure the bone mineral density (BMD g/cm2) to enable stratification into treatment strands and predict and prevent future fragility fractures.
Disease Severity | 2029
  Biochemical biomarkers (PARC/CCL18 ng/ml and Chitotriosidase umol/L/h) will be used to perform decease severity and follow-up response to treatment.
Bone Marrow Involvement | 2029
  MRI will allow us to assess the extent of Bone Marrow involvement and thus response to treatment by using the Bone Marrow Burden Score (BMB). The BMB is a semi quantitative MRI scoring system, using the sagittal T1 and T2 images of the lumbar spine and the coronal T1 and T2 of the femurs.
Bone avascular necrosis | 2029
  MRI will allow us to assess new avascular necrosis events (osteonecrosis).
Cognitive Function | 2019
  Frontal Assessment Battery (FAB) is used to assess early cognitive impairment in Type III patients and patients with diagnosis of Parkinson disease.
Cognitive Function | 2029
  Addenbrooke's Cognitive Examination - ACE-R and National Adult Reading Test are used in combinations to establish attention and orientation, memory, fluency, language and visuospatial orientation
Neurological Physical Assessment | 2029
  Modified Severity Scoring Tool (MSSt) is used to monitor neurological manifestations of NGD (Type III).
Multiple Myeloma | 2029
  Characterisation of new biomarkers in the peripheral blood mononuclear cells. (PBMCs), lipid analysis and Metabolomics screen.

SECONDARY OUTCOMES:
Quality of life and disease severity measures | 2029
  SF36; will be used to assess the patient reported quality of life. It is a generic measure of health status, as opposed to one that targets a specific age, disease, or treatment group. It has proven useful for conducting surveys of general and specific populations, comparing the relative burden of diseases, and differentiating the health benefits produced by a wide range of treatments.
Quality of life and disease severity measures | 2029
  EQ5D5L; the dimensions are (mobility, self care, usual activities, pain/discomfort, anxiety/depression). it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health. This tool will help facilitating the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions.
Quality of life and disease severity measures | 2029
  Hospital anxiety & depression scale (HADs); Assist researchers in detection of emotional disorder in patients under investigation and treatment
Quality of life and disease severity measures | 2029
  PedsQL (multidimensional fatigue scale); Enable researcher to assess if there is a link to level of patient reported fatigue and disease severity
Quality of life and disease severity measures | 2029
  PedsQL qual of life for paediatric ages. To assess participant reported quality of life.
Parkinson severity | 2029
  Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a clinical rating scale for Parkinson's disease (PD)
Biobank | 2020
  Biobank storage of historical and prospective human samples.
EyeSeeCam | 2029
  Objective quantifiable eye examination measuring eye movement

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Cox, MD, Principal Investigator — University of Cambridge
Locations (8):
- United Kingdom (8):
  - Birmingham Childrens Hospital, Birmingham
  - New Queen Elizabeth Hospital, Birmingham
  - Cambridge University Hospital, Cambridge
  - Great Ormond Street Hospital, London
  - National Hospital for Neurology and Neurosurgery, London
  - Royal Free Hospital, London
  - Royal Manchester Childrens Hospital, Manchester
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Yes
A Data sharing policy will be developed at the end of the study. Researchers will be able to make ethically approved requests to the Data owners for specific data (a charge will be made). What data sets will be available has yet to be decided by the Gaucherite Consortium Group.
Supporting Information: Study Protocol, ICF
Time Frame: At completion of study: however given the value of this cohort, efforts will be made to ensure permanence within the National Health Service and the context of NIHR.
Access Criteria: Individual applications made to Data Monitoring Committee and appropriate guarantees of confidentiality and ethical approval.

REFERENCES:
- [Background] D'Amore S, Page K, Donald A, Taiyari K, Tom B, Deegan P, Tan CY, Poole K, Jones SA, Mehta A, Hughes D, Sharma R, Lachmann RH, Chakrapani A, Geberhiwot T, Santra S, Banka S, Cox TM; MRC GAUCHERITE Consortium. In-depth phenotyping for clinical stratification of Gaucher disease. Orphanet J Rare Dis. 2021 Oct 14;16(1):431. doi: 10.1186/s13023-021-02034-6. PMID 34649574
- [Background] Donald A, Bjorkvall CK, Vellodi A; GAUCHERITE Consortium; Cox TM, Hughes D, Jones SA, Wynn R, Machaczka M. Thirty-year clinical outcomes after haematopoietic stem cell transplantation in neuronopathic Gaucher disease. Orphanet J Rare Dis. 2022 Jun 18;17(1):234. doi: 10.1186/s13023-022-02378-7. PMID 35717194
- [Background] Donald A, Tan CY, Chakrapani A, Hughes DA, Sharma R, Cole D, Bardins S, Gorges M, Jones SA, Schneider E. Eye movement biomarkers allow for the definition of phenotypes in Gaucher Disease. Orphanet J Rare Dis. 2020 Dec 17;15(1):349. doi: 10.1186/s13023-020-01637-9. PMID 33334373
- [Background] Adusumilli G, Kaggie JD, D'Amore S, Cox TM, Deegan P, MacKay JW, McDonald S; GAUCHERITE Consortium. Improving the quantitative classification of Erlenmeyer flask deformities. Skeletal Radiol. 2021 Feb;50(2):361-369. doi: 10.1007/s00256-020-03561-2. Epub 2020 Jul 30. PMID 32734372
- [Background] Yu B, Whitmarsh T, Riede P, McDonald S, Kaggie JD, Cox TM, Poole KES, Deegan P; MRC Gaucherite consortium. Deep learning-based quantification of osteonecrosis using magnetic resonance images in Gaucher disease. Bone. 2024 Sep;186:117142. doi: 10.1016/j.bone.2024.117142. Epub 2024 Jun 2. PMID 38834102
- [Derived] Donald A, Jones SA, Hughes DA, Church HJ; GAUCHERITE Consortium; Cox TM. Gaucher disease type 3: Classification of the chronic neuronopathic variant informed by genotype in a phenotypically diverse cohort. Genet Med. 2025 Sep;27(9):101502. doi: 10.1016/j.gim.2025.101502. Epub 2025 Jun 18. PMID 40542647
- [Derived] D'Amore S, Sano H, Chappell DDG, Chiarugi D, Baker O, Page K, Ramaswami U, Johannesdottir F, Cox TM, Deegan P, Poole KE; MRC Gaucherite Consortium; MRC Gaucherite Consortium Collaborators. Radiographic Cortical Thickness Index Predicts Fragility Fracture in Gaucher Disease. Radiology. 2023 Apr;307(1):e212779. doi: 10.1148/radiol.212779. Epub 2022 Dec 20. PMID 36537898